CLINICAL TRIAL: NCT03128892
Title: Oxygen Reserve Index Validation for RD Lite Sensors
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP18600A-135_197
Record Dates: First submitted 2017-04-14; First posted 2017-04-25 (Actual); Results first posted 2020-07-23 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects are enrolled into the test group and all subjects received the Noninvasive Oxygen Reserve Index - RD Lite Sensors
  Interventions: Device: Oxygen Reserve Index - RD Lite Sensors

INTERVENTIONS:
Device: Oxygen Reserve Index - RD Lite Sensors

SUMMARY:
Oxygen Reserve Index (ORI) is a parameter that provides information on arterial partial pressure of oxygen (PaO2). In this study, the PaO2 is varied by controlling the concentration of oxygen the study volunteer breathes. The ORI device measurement is analyzed by comparing it to the PaO2 measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Competent non-smoking (smokers including e-cigarette users) adults between the ages of 18 and 50 years of age.
* We may also be interested in specifically recruiting smokers for some portions of this study as well as non-smokers for other portions of this study.
* Must weigh a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* BMI less than or equal to 35
* Must have a hemoglobin value greater than or equal to 11 g/dL.
* Baseline heart rate > 45 bpm and < 85 bpm.
* CO value less than or equal to 2.0% FCOHb (unless we are specifically interested in recruiting smokers)
* Physical status of ASA I or II (American Society of Anesthesiology Class 1; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease)
* Blood Pressure (Systolic BP less than for equal to 140 mmHg and Diastolic BP less than or equal to 90 mmHg).
* Able to read and communicate in English
* Has signed written informed consent
* Female, non-pregnant.
* Female subjects will be provided with a pregnancy test free of charge.

Exclusion Criteria:

* Subjects who do not understand the study and the risks involved.
* Subjects with open wounds, lacerations, inflamed tattoos or piercings, visible healing wounds.
* Subjects with frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse. Subjects who uses recreational drugs.
* Subject has experienced a head injury with loss of consciousness within the last year.
* Any chronic bleeding disorders (i.e. hemophilia)
* Any history of a stroke, myocardial infarction, seizures or heart attack.
* Any cancer or history of cancer (not including skin cancer).
* Chronic neurological diseases (i.e. multiple sclerosis, Huntington's Disease).
* Any cardiac dysrhythmias (i.e. atrial fibrillation)(without physicians clearance)
* Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subjects' level of consciousness.
* Known or concurrent chronic usage of psychoactive or anticonvulsive drugs. Subjects with psychiatric conditions or are on psychiatric medications (i.e. tricyclic antidepressants, MAO inhibitors, Lithium, neuroleptics, anxiolytics or antipsychotics, except SSRIs).
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study, such as Reynauds Syndrome.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome
* Inability to tolerate sitting still or maintain minimal movement for up to 90 minutes.
* For studies involving finger sensors: subjects with polished, gel or acrylic nails, skin abnormalities affecting the fingers or arms (such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection), distinct finger edema, substantial skin breakdown damaged and/or finger nail deformities (specific finger will not be used, unless we are specifically testing sensors in use with nail polish, gel, and /or acrylic nails).
* Subjects who have/are currently taking anticoagulant medication.
* Subjects who have had caffeine consumption the day of the study.
* Subjects who have taken pain medication within 24 hours of start of study. Unless minimal preventative dose recommended for adults (discretion of physician).
* Subjects having either signs or history of peripheral ischemia.
* Subjects who have had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, Urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subjects who have had minor surgery or conditions in the past two months including but not limited to minor foot surgery (bunion), arthroscopic procedure, blood donation, plasma donation, skin biopsy/ procedures, root canal, fractures, eye surgery, and other minor procedures.
* Subjects that have been on antibiotics had congestion, head colds, flu, ear infection, chest congestion will have a 2 week waiting period from the time of finishing medications and must have no more symptoms.
* Subjects with claustrophobia, or anxiety.
* Subjects who have been in severe car accidents or a similar type of accidents will have a 12 month waiting period, from the time of the accident; unless upon further medical history questions the physician determines it does not place the subject in any additional harm, increase their risk, or compromise the subjects' safety.
* Subjects who have had a concussion will have a 12 month waiting period, from the time of the concussion.
* Subjects with chronic unresolved asthma, lung disease or respiratory disease.
* Subjects with allergies to lidocaine, latex, adhesives, or plastic.
* Subjects with heart conditions, Diabetes or hypertension.
* Subjects who have given vaginal delivery will have a 6 month waiting period. Subjects who had a pregnancy terminated, a miscarriage or had a C-section will have a 12 month waiting period.
* Subjects who intend on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study involving an arterial blood draw and/or arterial line placement.
* Discretion of investigator/study staff

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygen Reserve Index (ORi) - RD Lite Sensors: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Oxygen Reserve Index - RD Lite Sensors.
Period: Overall Study
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
Started | 34
Completed | 31
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 12
  Asian or Pacific Islander | 1
  Caucasian | 5
  Hispanic | 13
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Specificity of ORI to Detect Drops in Oxygenation
Description: A measure of the ORI parameter's ability to detect changes in dissolved oxygen levels in blood plasma. Specificity, as measured in this outcome, is the probability of ORI not dropping when there is no drop in blood oxygen levels (desaturation).
Time Frame: 1-5 hours per subject
Measure: Number; unit: percentage of true negative
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
Number analyzed (Participants) | 31
percentage of true negative
  PaO2 Threshold: 110 mmHg | 98.50
  PaO2 Threshold: 120 mmHg | 96.68
  PaO2 Threshold: 130 mmHg | 98.89
  PaO2 Threshold: 140 mmHg | 96.95
  PaO2 Threshold: 150 mmHg | 97.67
  PaO2 Threshold: 160 mmHg | 94.75
  PaO2 Threshold: 170 mmHg | 93.60
  PaO2 Threshold: 180 mmHg | 96.23
  PaO2 Threshold: 190 mmHg | 95.82

2. Primary Outcome: Sensitivity of ORI to Detect Drops in Oxygenation
Description: A measure of the ORI parameter's ability to detect changes in dissolved oxygen levels in blood plasma. Sensitivity, as measured in this outcome, is the probability of ORI dropping when there is a drop in blood oxygenation levels (desaturation).
Time Frame: 1-5 hours
Measure: Number; unit: percentage of true positives
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
Number analyzed (Participants) | 31
percentage of true positives
  PaO2 Threshold: 110 mmHg | 84.96
  PaO2 Threshold: 120 mmHg | 89.85
  PaO2 Threshold: 130 mmHg | 85.51
  PaO2 Threshold: 140 mmHg | 89.47
  PaO2 Threshold: 150 mmHg | 86.17
  PaO2 Threshold: 160 mmHg | 87.13
  PaO2 Threshold: 170 mmHg | 83.96
  PaO2 Threshold: 180 mmHg | 85.40
  PaO2 Threshold: 190 mmHg | 88.27

3. Primary Outcome: Concordance of ORI to Detect Drops in Oxygenation
Description: A measure of the ORI parameter's ability to detect changes in dissolved oxygen levels in blood plasma. Concordance, as measured in this outcome, is the probability of ORI to respond accurately to changes (or lack of thereof) in underlying blood oxygenation levels. It is computed as a ratio of true classifications (true positives and true negatives) to the sample size. An ideal detector will have a concordance value of 1 (or 100%).
Time Frame: 1-5 hours
Measure: Number; unit: percentage of accuracy
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
Number analyzed (Participants) | 31
percentage of accuracy
  PaO2 Threshold: 110 mmHg | 88.83
  PaO2 Threshold: 120 mmHg | 92.46
  PaO2 Threshold: 130 mmHg | 91.47
  PaO2 Threshold: 140 mmHg | 93.33
  PaO2 Threshold: 150 mmHg | 93.00
  PaO2 Threshold: 160 mmHg | 92.16
  PaO2 Threshold: 170 mmHg | 90.80
  PaO2 Threshold: 180 mmHg | 93.78
  PaO2 Threshold: 190 mmHg | 94.39

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | Oxygen Reserve Index (ORi) - RD Lite Sensors
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxygen Reserve Index (ORi) - RD Lite Sensors (N=34)
Arterial line site sensitivity (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03128892/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03128892/SAP_001.pdf